CLINICAL TRIAL: NCT00846742
Title: Reduced Duration Stanford V Chemotherapy With or Without Low-Dose Tailored-Field Radiation Therapy For Favorable Risk Pediatric Hodgkin Lymphoma
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Young Patients With Favorable-Risk Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOD08; NCI-2009-01138 (Registry Identifier: NCI's Clinical Trial Reporting Program)
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants receive Stanford V Chemotherapy with or without radiation therapy. Patients receive doxorubicin hydrochloride IV and vinblastine IV on day 1 of weeks 1, 3, 5, and 7; mechlorethamine hydrochloride IV on day 1 of weeks 1 and 5; vincristine sulfate IV and bleomycin IV on day 1 of weeks 2, 4, 6, and 8; etoposide IV on day 1 of weeks 3 and 7; and prednisone orally (PO) three times daily every other day of weeks 1-8. Beginning 2-3 weeks after completion of chemotherapy, patients not achieving complete response undergo radiation therapy to individual nodal sites (tailored fields)
  Interventions: Drug: Stanford V Chemotherapy; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Stanford V Chemotherapy — The Stanford V regimen is an abbreviated, multi-agent, dose-intensive regimen that utilizes many of the most active chemotherapy agents for Hodgkin lymphoma: Vinblastine, Doxorubicin, Vincristine, Bleomycin, Mechlorethamine, Etoposide, and Prednisone
Radiation: Radiation Therapy — Patients who achieve less than a complete response after 8 weeks of chemotherapy will receive 25.5 Gy to individual nodal sites (tailored fields) starting 2-3 weeks following completion of all chemotherapy and recovery of ANC to at least 1000.

SUMMARY:
This phase II trial is studying how well combination chemotherapy with or without radiation therapy works in treating young patients with favorable-risk Hodgkin lymphoma. Drugs used in chemotherapy, such as doxorubicin hydrochloride, vinblastine, mechlorethamine hydrochloride, vincristine sulfate, bleomycin, etoposide, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Radiation therapy uses high-energy x-rays to kill cancer cells for those patients that still had residual cancer at the end of chemotherapy. Giving combination chemotherapy with radiation therapy may kill more cancer cells and allow doctors to save the part of the body where the cancer started.

DETAILED DESCRIPTION:
Patients receive doxorubicin hydrochloride intravenously (IV) and vinblastine IV on day 1 of weeks 1, 3, 5, and 7; mechlorethamine hydrochloride IV on day 1 of weeks 1 and 5; vincristine sulfate IV and bleomycin IV on day 1 of weeks 2, 4, 6, and 8; etoposide IV on day 1 of weeks 3 and 7; and prednisone orally (PO) three times daily every other day for 8 weeks. Two to 3 weeks after all chemotherapy is given, patients not achieving a complete response undergo radiation therapy to individual nodal sites (tailored fields).

PRIMARY OBJECTIVES:

1. To increase the complete response rate of favorable risk patients (excluding all patients with stage IA nodular lymphocyte predominant Hodgkin lymphoma) after 8 weeks Stanford V by at least 20% compared to favorable risk patients on HOD 99 after 8 weeks vincristine, doxorubicin hydrochloride, methotrexate and prednisone (VAMP).

SECONDARY OBJECTIVES:

1. To estimate the disease failure rate within the radiation fields.
2. To examine patterns of treatment failure for children treated with low dose tailored field radiation therapy.
3. To describe acute hematologic and infectious toxicities as they relate to transfusion requirements, growth factor support, episodes of febrile neutropenia, and hospitalizations, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
4. To compare the survival distributions (event-free and overall) and cumulative incidence of local failure and toxicities of favorable risk patients treated with 8 weeks of Stanford V chemotherapy and low-dose tailored-field radiation to those on the favorable risk group of the HOD 99 study that received VAMP and low-dose involved-field radiation.
5. To compare the survival distributions between patients that will not be prescribed radiotherapy after 8 weeks Stanford V and those patients on HOD 99 that did not receive radiotherapy after VAMP.
6. To estimate the event-free survival distributions of favorable risk patients treated with Stanford V chemotherapy alone and patients treated with Stanford V chemotherapy plus low dose tailored field radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, previously untreated Hodgkin lymphoma.
* Age: Participants must be 21 years of age or younger
* Stage must be classified as one of the following:

Ann Arbor stage IA or IIA with:

* Non-bulky mediastinal disease (< 33% mediastinal to thoracic ratio on CXR)
* < 3 nodal regions involved on the same side of the diaphragm
* No "E" lesion
* Female patients who are post-menarchal must have a negative pregnancy test. Patients of reproductive potential must agree to use an effective contraceptive method.
* Signed informed consent
* If re-evaluation of a patient's disease shows intermediate risk features, the patient will be removed from the HOD08.

Exclusion Criteria:

* Intermediate or High risk disease, defined as Stage IB, any III or IV or IA/IIA with "E" lesion(s), 3 or more nodal sites involved, or bulky mediastinal adenopathy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2009-06-05 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2028-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Ehrhardt, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (6):
- United States (6):
  - Packard Children's Hospital, Stanford University, Palo Alto, California
  - Rady Children's Hospital- San Diego, San Diego, California
  - Children's Hospital of Illinois at OSF St. Francis Medical Center, Peoria, Illinois
  - Maine Children's Cancer Program (MCCP), Scarborough, Maine
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Flerlage JE, Feraco AM MD, MMSc, Zhou Y, Zheng Y MS, Liang J, Lucas JT Jr, Friedmann AM, Weinstein HJ, Yock TI, Shulkin BL, Kaste SC, Marks LJ, Ehrhardt MJ, Dixon SB, Howard S, de Alarcon P, Luna-Fineman S, Geddis AE, Larsen EC, Marcus KJ, Billett A, Donaldson SS, Hudson MM, Metzger ML, Krasin MJ, Link MP. Dose-dense chemotherapy enables elimination of RT for majority of low-risk pediatric Hodgkin lymphoma: PHC study HOD08. Blood. 2026 Jan 13:blood.2025029535. doi: 10.1182/blood.2025029535. Online ahead of print. PMID 41529162
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 88 participants were enrolled from 5 institutions between June 2009 and October 2018.
Pre-assignment Details: Two out of 88 enrolled patients are ineligible and were removed from the study. They were determined to be intermediate risk rather than low risk. One was taken off study after being re-consented on an expired consent and treated with cyclophosphamide instead of mechlorethamine; 1 patient withdrew from study but was evaluable for primary objective.
Groups:
- Stanford V Chemotherapy: Ann Arbor stage IA or IIA with:
  1. Non-bulky mediastinal disease (<33% mediastinal to thoracic ratio on chest x-ray)
  2. < 3 nodal regions involved on the same side of the diaphragm
  3. No extranodal extension of disease
Period: Overall Study
Arm/Group | Stanford V Chemotherapy
Started | 85
With Radiation Therapy (RT) (Seventeen (17) participants out of the 85 analyzed received radiation therapy (RT)) | 17
Without Radiation Therapy (RT) (Sixty-eight (68) participants out of the 85 analyzed did not receive RT) | 68
Completed | 84
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 66
  Race: Black | 8
  Race: Asian | 3
  Race: Multiple Race (NOS) | 3
  Race: Other | 3
  Race: American Ind / Alaskan / White | 1
  Race: Asian and White | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States: St. Jude Children's Research Hospital | 46
  United States: Stanford University Medical Center | 15
  United States: Dana Farber Cancer Institute | 13
  United States: Rady Children's Hospital San Diego | 6
  United States: Maine Medical Center | 5
Stage: IA, IIA [Count of Participants; unit: Participants] — Stages were according to the Ann Arbor Classification (stage I: one single lymph node group involved, stage II: 2 lymph node groups involved on one side of the diaphragm). "A" stands for absence of "B" symptoms (fevers, night sweats or weight loss).
  Participants
    IA | 29
    IIA | 56

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate Estimate
Description: To increase the complete response rate of favorable risk patients (excluding all patients with stage IA nodular lymphocyte predominant Hodgkin lymphoma) after 8 weeks Stanford V by at least 20% compared to favorable risk patients on HOD 99 after 8 weeks VAMP (NCT number: NCT00145600) .Complete response definition: Disappearance of all measurable or evaluable disease, signs, symptoms and biochemical changes related to the tumor. Biopsy confirmation is not mandatory. Residual PET-negative CT scan abnormalities representing > 75% reduction (as measured by the product of 2 perpendicular diameters of lesions by CT or MR imaging) in the original tumor volume will be considered scar tissue without active tumor.
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Stanford V Chemotherapy: Non-stage IA non-LP favorable risk participants receive 8 weeks of Stanford V chemotherapy.
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 56
percentage of participants | 77 [64 to 87]
Statistical Analysis 1: Comparison: Stanford V Chemotherapy; The proportion of patients' complete response rate was provided with a 95% confidence interval; Test type: Superiority; p = 0.0003, Exact Binominal Test — Comparison of proportion of patients' complete response rate between HOD99 (NCT number: NCT00145600) and HOD08

2. Secondary Outcome: Acute Hematologic Toxicities
Description: Description of acute hematologic toxicities as they relate to transfusion requirements, growth factor support, episodes of febrile neutropenia and hospitalizations, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. The acute hematologic toxicities were summarized descriptively.
Time Frame: 6 months
Measure: Number; unit: adverse events
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 85
adverse events
  Neutrophils/granulocytes (ANC/AGC) | 64
  Leukocytes (total WBC) | 74
  Lymphopenia | 54
  Hemoglobin | 14
  Platelets | 1

3. Secondary Outcome: Acute Infectious Toxicities
Description: Description of acute infectious toxicities as they relate to transfusion requirements, growth factor support, episodes of febrile neutropenia and hospitalizations, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. The acute infectious toxicities were summarized descriptively.
Time Frame: 6 months
Measure: Number; unit: Adverse events
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 85
Adverse events
  Febrile neutropenia | 8
  Infection, Blood | 2
  Infection, Upper Airway NOS | 1

4. Secondary Outcome: Disease Failure Rate Within Radiation Fields
Description: Defined as disease that recurs in the initially involved nodal region within the field of irradiation. The disease failure rate within the radiation fields will be estimated with a 95% confidence interval using appropriate methods (e.g., estimate cumulative incidence in the presence of competing risks).
Time Frame: median 2 year post therapy
Measure: Number (95% Confidence Interval); unit: probability that the event occurs
Groups:
- With Radiation Therapy: Favorable Risk Patients Treated with Stanford V Chemotherapy Plus Low Dose Tailored-field Radiation
Arm/Group | With Radiation Therapy
Number analyzed (Participants) | 17
probability that the event occurs | 0.059 [0.003 to 0.242]

5. Secondary Outcome: Treatment Failure Patterns for Children Treated With Tailored-field Radiation
Description: Descriptive statistics related to local/distant failure will be produced. The cumulative incidence of local failure will be estimated and effects of prognostic factors will be examined. Effect of competing risks (distant failure, second malignancy and death) will be taken into account. Relapse rate within the radiation fields will be estimated and confidence interval will also be calculated.
Time Frame: median 2 years post therapy
Measure: Number (95% Confidence Interval); unit: probability that the event occurs
Groups:
- With Radiation Therapy (RT): Favorable Risk Patients Treated with Stanford V Chemotherapy Plus Low Dose Tailored-field Radiation
Arm/Group | With Radiation Therapy (RT)
Number analyzed (Participants) | 17
probability that the event occurs
  2-year Cumulative incidence of distant failure | 0.000 [0.000 to 0.000]
  2-year Cumulative incidence of local failure | 0.059 [0.003 to 0.242]

6. Secondary Outcome: Prognostic Factors for Local Failure in Children Treated With Tailored-Field Radiation: Age
Description: Age was examined for the association with cumulative incidence of local failure. Effect of competing risks (distant failure, second malignancy and death) will be taken into account. Fine and Gray's competing risk regression model with Wald test will be used to compute the p value for the statistical significance.
Time Frame: median 2 years post therapy
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | With Radiation Therapy (RT)
Number analyzed (Participants) | 17
hazard ratio | 0.969 [0.810 to 1.159]
Statistical Analysis 1: Comparison: With Radiation Therapy (RT); Test type: Superiority; p = 0.732, Fine-Gray model; Hazard Ratio (HR) = 0.969, 95% CI 2-sided [0.810 to 1.159] — The sub-distribution hazard ratio for the 2-year cumulative incidence of local failure with a 1-year increase in age

7. Secondary Outcome: Prognostic Factors for Local Failure in Children Treated With Tailored-Field Radiation: Gender
Description: Gender was examined for the association with cumulative incidence of local failure. Effect of competing risks (distant failure, second malignancy and death) will be taken into account. Fine and Gray's competing risk regression model with Wald test will be used to compute the p value for the statistical significance.
Time Frame: median 2 years post therapy
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | With Radiation Therapy (RT)
Number analyzed (Participants) | 17
hazard ratio | 0.000 [0.000 to 0.000]
Statistical Analysis 1: Comparison: With Radiation Therapy (RT); Male vs. Female, with Female as the reference level; Test type: Superiority; p < 0.001, Fine-Gray model; Hazard Ratio (HR) = 0.000, 95% CI 2-sided [0.000 to 0.000] — The sub-distribution hazard ratio for the 2-year cumulative incidence of local failure comparing males to females

8. Secondary Outcome: Prognostic Factors for Local Failure in Children Treated With Tailored-Field Radiation: Stage
Description: Stage was examined for the association with cumulative incidence of local failure. Effect of competing risks (distant failure, second malignancy and death) will be taken into account. Fine and Gray's competing risk regression model with Wald test will be used to compute the p value for the statistical significance.
Time Frame: median 2 years post therapy
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | With Radiation Therapy (RT)
Number analyzed (Participants) | 17
hazard ratio | 30101.410 [3329.573 to 272135.500]
Statistical Analysis 1: Comparison: With Radiation Therapy (RT); Stage IIA vs. Stage IA, with Stage IA as the reference level; Test type: Superiority; p < 0.001, Fine-Gray model; Hazard Ratio (HR) = 30101.410, 95% CI 2-sided [3329.573 to 272135.500] — The sub-distribution hazard ratio for the 2-year cumulative incidence of local failure comparing Stage IIA to Stage IA

9. Secondary Outcome: Prognostic Factors for Local Failure in Children Treated With Tailored-Field Radiation: Histology
Description: Histology was examined for its association with the cumulative incidence of local failure. Effect of competing risks (distant failure, second malignancy and death) will be taken into account. Fine and Gray's competing risk regression model with the Wald test will be used to compute the p-value for statistical significance.
Time Frame: median 2 years post therapy
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | With Radiation Therapy (RT)
Number analyzed (Participants) | 17
hazard ratio | 34027.680 [4072.872 to 284291.600]
Statistical Analysis 1: Comparison: With Radiation Therapy (RT); Classical (all combined) vs. Nodular lymphocyte predominant, with Nodular lymphocyte predominant as the reference level; Test type: Superiority; p < 0.001, Fine-Gray model; Hazard Ratio (HR) = 34027.680, 95% CI 2-sided [4072.872 to 284291.600] — The sub-distribution hazard ratio for the 2-year cumulative incidence of local failure comparing Classical (all combined) to Nodular Lymphocyte Predominant Hodgkin Lymphoma

10. Secondary Outcome: Comparison of Event-free and Overall Survival Distributions, and Cumulative Incidence of Local Failure of Patients Treated on This Study to Outcome in the Favorable Risk Group of HOD99
Description: Log-rank tests are used to compare event-free survival and overall survival. Event-free survival is defined as time interval from the date of study enrollment to the date of first event (relapsed or progressive disease, second malignancy, or death from any cause) or to last follow-up for patients without events. Survival is defined as time interval from study enrollment to date of death from any cause or to date of last follow-up. Gray's test used to compare cumulative incidence of local failure between favorable risk patients treated on this protocol vs. treated on HOD99 and other regimens.
Time Frame: median 2 years post therapy
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- HOD08 Participants: Ann Arbor stage IA or IIA with:
  1. Non-bulky mediastinal disease (<33% mediastinal to thoracic ratio on chest x-ray)
  2. < 3 nodal regions involved on the same side of the diaphragm
  3. No extranodal extension of disease
- HOD99 Participants: Favorable Risk participants treated on the earlier HOD99 protocol (NCT00145600) at St. Jude Children's Research Hospital.
Arm/Group | HOD08 Participants | HOD99 Participants
Number analyzed (Participants) | 85 | 88
probability
  2-year Event-free Survival (EFS) Probability | 0.939 [0.889 to 0.992] | 0.909 [0.851 to 0.971]
  2-year Overall Survival (OS) Probability | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  2-year Cumulative Incidence (CI) of Local Failure | 0.061 [0.022 to 0.127] | 0.068 [0.028 to 0.134]
Statistical Analysis 1: Comparison: HOD08 Participants vs HOD99 Participants; Comparing the 2-year EFS between HOD08 Participants and HOD99 Participants; Test type: Superiority; p = 0.461, Log Rank
Statistical Analysis 2: Comparison: HOD08 Participants vs HOD99 Participants; Comparing the 2-year OS between HOD08 Participants and HOD99 Participants; Test type: Superiority; p = 1.000, Log Rank
Statistical Analysis 3: Comparison: HOD08 Participants vs HOD99 Participants; Comparing the 2-year CI of Local Failure between HOD08 Participants and HOD99 Participants; Test type: Superiority; p = 0.836, Gray's test

11. Secondary Outcome: Comparison of Toxicities of Patients Treated on This Study to Outcome and Toxicities in the Favorable Risk Group of HOD99
Description: Comparison of the toxicities with grade > 2 of low-risk patients treated with reduced duration Stanford V chemotherapy with or without low-dose tailored-field radiation (current HOD08 protocol) to those of favorable-risk patients on HOD99 (NCT00145600). Grading of toxicities for HOD08 and HOD99 used the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: median 2 years post therapy
Population: Additional description can be found here for the following Row Titles:
  Febrile neutropenia - (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
  Infection, Blood - (documented clinically or microbiologically documented infection) (ANC<1.0x10^9/L, fever > 38.5C)
  Infection, Paranasal - (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Measure: Number; unit: adverse events
Groups:
- HOD08 - Grade 3; HOD08 - Grade 4; HOD08 - Grade 5: Participants in current study.
- HOD99 - Grade 3; HOD99 - Grade 4; HOD99 - Grade 5: Favorable Risk participants treated on the earlier HOD99 protocol (NCT00145600) at St. Jude Children's Research Hospital.
Arm/Group | HOD08 - Grade 3 | HOD08 - Grade 4 | HOD08 - Grade 5 | HOD99 - Grade 3 | HOD99 - Grade 4 | HOD99 - Grade 5
Number analyzed (Participants) | 85 | 85 | 85 | 88 | 88 | 88
adverse events
  ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 0 | 0 | 2 | 0 | 0
  AST, SGOT(serum glutamic oxaloacetic transaminase) | 0 | 0 | 0 | 2 | 0 | 0
  Bicarbonate, serum-low | 0 | 0 | 0 | 0 | 1 | 0
  Blood/Bone Marrow - Other (Specify, __) | 0 | 0 | 0 | 0 | 1 | 0
  Calcium, serum-low (hypocalcemia) | 0 | 0 | 0 | 0 | 1 | 0
  Constipation | 1 | 0 | 0 | 1 | 0 | 0
  Dehydration | 1 | 0 | 0 | 1 | 0 | 0
  Febrile neutropenia | 4 | 2 | 0 | 1 | 1 | 0
  Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) | 0 | 0 | 0 | 2 | 0 | 0
  Flu-like syndrome | 1 | 0 | 0 | 0 | 0 | 0
  Gastritis (including bile reflux gastritis) | 0 | 0 | 0 | 1 | 0 | 0
  Glucose, serum-high (hyperglycemia) | 0 | 0 | 0 | 1 | 1 | 0
  Hemoglobin | 6 | 2 | 0 | 1 | 0 | 0
  Hypotension | 1 | 0 | 0 | 0 | 0 | 0
  Hypoxia | 1 | 0 | 0 | 0 | 0 | 0
  Infection, Blood | 0 | 0 | 0 | 1 | 0 | 0
  Infection, Paranasal | 0 | 0 | 0 | 1 | 0 | 0
  Infection with normal ANC or Grade 1 or 2 neutrophils, Blood | 2 | 0 | 0 | 1 | 0 | 0
  Infection with normal ANC or Grade 1 or 2 neutrophils, Catheter-related | 0 | 0 | 0 | 1 | 0 | 0
  Infection with normal ANC or Grade 1 or 2 neutrophils, Pharynx | 0 | 0 | 0 | 1 | 0 | 0
  Infection with normal ANC or Grade 1 or 2 neutrophils, Skin (cellulitis) | 0 | 0 | 0 | 1 | 0 | 0
  Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS | 1 | 0 | 0 | 0 | 0 | 0
  Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS | 1 | 0 | 0 | 1 | 0 | 0
  Infection with unknown ANC, Lung (pneumonia) | 0 | 0 | 0 | 1 | 0 | 0
  Insomnia | 0 | 0 | 0 | 1 | 0 | 0
  Leukocytes (total WBC) | 34 | 18 | 0 | 23 | 0 | 0
  Lymphopenia | 23 | 10 | 0 | 0 | 0 | 0
  Magnesium, serum-high (hypermagnesemia) | 1 | 0 | 0 | 0 | 0 | 0
  Magnesium, serum-low (hypomagnesemia) | 0 | 0 | 0 | 0 | 1 | 0
  Mood alteration, Depression | 0 | 0 | 0 | 3 | 0 | 0
  Nausea | 1 | 0 | 0 | 0 | 0 | 0
  Neuropathy: sensory | 0 | 0 | 0 | 4 | 0 | 0
  Neutrophils/granulocytes (ANC/AGC) | 32 | 25 | 0 | 36 | 51 | 0
  Obstruction, GU, Bladder | 1 | 0 | 0 | 0 | 0 | 0
  Pain - Other (Specify, __) | 1 | 0 | 0 | 0 | 0 | 0
  Pain, Abdomen NOS | 2 | 0 | 0 | 0 | 0 | 0
  Pain, Bone | 0 | 0 | 0 | 1 | 1 | 0
  Pain, Chest/thorax NOS | 0 | 1 | 0 | 0 | 0 | 0
  Pain, Extremity-limb | 1 | 0 | 0 | 0 | 0 | 0
  Pain, Joint | 0 | 0 | 0 | 2 | 0 | 0
  Pain, Neuralgia/peripheral nerve | 1 | 0 | 0 | 0 | 0 | 0
  Personality/behavioral | 0 | 0 | 0 | 1 | 0 | 0
  Phosphate, serum-low (hypophosphatemia) | 0 | 0 | 0 | 0 | 1 | 0
  Potassium, serum-high (hyperkalemia) | 0 | 1 | 0 | 0 | 0 | 0
  Potassium, serum-low (hypokalemia) | 0 | 0 | 0 | 1 | 1 | 0
  Renal failure | 1 | 0 | 0 | 0 | 0 | 0
  Sodium, serum-low (hyponatremia) | 0 | 0 | 0 | 0 | 1 | 0
  Thrombosis/embolism (vascular access-related) | 0 | 0 | 0 | 2 | 0 | 0
  Thrombosis/thrombus/embolism | 1 | 0 | 0 | 1 | 0 | 0
  Vomiting | 2 | 0 | 0 | 3 | 0 | 0
  Weight gain | 0 | 0 | 0 | 1 | 0 | 0

12. Secondary Outcome: Comparison of Event-free and Overall Survival Distributions and Cumulative Incidence of Local Failure Between Patients That Will Not be Prescribed Radiotherapy After 8 Weeks Stanford V and Those Patients on HOD99 That Received VAMP Without Radiotherapy
Description: Log-rank tests are used to compare event-free survival and overall survival. Event-free survival is defined as time interval from the date of study enrollment to the date of first event (relapsed or progressive disease, second malignancy, or death from any cause) or to last follow-up for patients without events. Survival is defined as time interval from study enrollment to date of death from any cause or to date of last follow-up. Gray's test used to compare cumulative incidence of local failure between favorable risk patients treated on this protocol vs. treated on HOD99 and other regimens. Patients who will not be prescribed Radiotherapy in both protocols are those who achieved CR on the response assessment after chemotherapy.
Time Frame: median 2 years post therapy
Population: HOD08 - CR: Participants who achieved CR after chemotherapy and were not prescribed RT. Two patients without RT were excluded: 1 was prescribed but did not receive it due to consent withdrawal, and 1 withdrew with no response results.
  HOD99 - CR: Favorable Risk participants from NCT00145600 (HOD99) who achieved CR after chemotherapy and were not prescribed RT. Two patients prescribed RT but not receiving it were excluded: 1 due to progressive disease and 1 due to consent withdrawal.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- HOD08 - CR: Participants in the current study who have achieved a "CR" (Complete Response) on Response Assessment after chemotherapy.
- HOD99 - CR: Favorable Risk participants treated on the earlier HOD99 protocol (NCT00145600) at St. Jude Children's Research Hospital who have achieved a 'CR' on Response Assessment after chemotherapy
Arm/Group | HOD08 - CR | HOD99 - CR
Number analyzed (Participants) | 66 | 47
probability
  2-year Event-free Survival (EFS) Probability | 0.938 [0.881 to 0.999] | 0.894 [0.810 to 0.986]
  2-year Overall Survival (OS) Probability | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000]
  2-year Cumulative Incidence (CI) of Local Failure | 0.062 [0.020 to 0.139] | 0.106 [0.039 to 0.214]
Statistical Analysis 1: Comparison: HOD08 - CR vs HOD99 - CR; Comparing the 2-year EFS between HOD08 - CR and HOD99 - CR; Test type: Superiority; p = 0.384, Log Rank
Statistical Analysis 2: Comparison: HOD08 - CR vs HOD99 - CR; Comparing the 2-year OS between HOD08 - CR and HOD99 - CR; Test type: Superiority; p = 1.000, Log Rank
Statistical Analysis 3: Comparison: HOD08 - CR vs HOD99 - CR; Comparing the 2-year CI of Local Failure between HOD08 - CR and HOD99 - CR; Test type: Superiority; p = 0.386, Gray's test

13. Secondary Outcome: Event-free Survival Distributions of Favorable Risk Patients Treated With Stanford V Chemotherapy Alone and Patients Treated With Stanford V Chemotherapy Plus Low Dose Tailored-field Radiation
Description: Event-free survival distributions of favorable risk patients treated with Stanford V chemotherapy alone and patients treated with Stanford V chemotherapy plus low dose tailored field radiation will be estimated by the Kaplan-Meier method.
Time Frame: median 2 years post therapy
Population: Stanford V Chemotherapy Alone: Out of the 68 patients treated with Stanford V chemotherapy alone, without low-dose tailored-field radiation:
  66 patients were not prescribed radiotherapy as they achieved a Complete Response (CR) on the Response Assessment after chemotherapy.
  One patient didn't achieve a CR but withdrew from the study before receiving radiotherapy.
  One patient had a missing response result and withdrew from the study without undergoing radiotherapy.
Measure: Number (95% Confidence Interval); unit: probability of event free survival
Groups:
- Stanford V Chemotherapy Alone: Favorable Risk Patients Treated with Stanford V Chemotherapy Alone without Low Dose Tailored-field Radiation
Arm/Group | Stanford V Chemotherapy Alone | With Radiation Therapy (RT)
Number analyzed (Participants) | 68 | 17
probability of event free survival | 0.939 [0.882 to 0.999] | 0.941 [0.836 to 1.000]
Statistical Analysis 1: Comparison: Stanford V Chemotherapy Alone vs With Radiation Therapy (RT); Comparing the 2-year EFS of patients treated without and with RT; Test type: Superiority; p = 0.986, Log Rank

ADVERSE EVENTS:
Time Frame: Acute adverse events were collected from study enrollment up to 4 weeks after completion of chemotherapy/radiation therapy, whichever came last. Long term toxicity was captured at every visit up to 5 years from study enrollment.
Arm/Group | Stanford V Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/85
Serious Adverse Events (participants affected / at risk) | 1/85
Other Adverse Events (participants affected / at risk) | 58/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanford V Chemotherapy (N=85)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanford V Chemotherapy (N=85)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 39 (63)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 36 (73)
Lymphopenia (Blood and lymphatic system disorders) | 22 (54)
Hemoglobin (Blood and lymphatic system disorders) | 9 (14)
Febrile neutropenia (Infections and infestations) | 6 (8) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever ≥38.5°C)

LIMITATIONS AND CAVEATS:
During a mechlorethamine shortage cyclophosphamide was administered instead leading to inferior outcome in intermediate and high risk patients. These patients were replaced in this protocol. The study was closed early after our new protocol opened. Enrolled participants may be followed for 10 years after completion of therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT00846742/Prot_SAP_002.pdf